CLINICAL TRIAL: NCT01452724
Title: A Phase 3, Randomized, Double Blind, Double-Dummy, Multicenter, Parallel Group Comparison Study to on Efficacy and Safety of Oral Once-Daily Administration of TAK-438 20 mg Comparing With AG-1749 in Patients With Duodenal Ulcer
Brief Title: Efficacy and Safety of TAK-438 Compared to AG-1749 (Lansoprazole) in the Treatment of Duodenal Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CCT-102; U1111-1123-8648 (Registry Identifier: WHO); JapicCTI-111608 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-16; First posted 2011-10-17 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Duodenal Ulcer
Keywords: Drug Therapy
MeSH Terms: conditions — Duodenal Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438; Drug: Placebo
- Lansoprazole 30 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole; Drug: Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 20 mg, tablets, orally, once daily for up to 6 weeks.
  Arms: TAK-438 20 mg QD
Drug: Placebo — Lansoprazole placebo-matching capsules, orally, once daily for up to 6 weeks.
  Arms: TAK-438 20 mg QD
Drug: Lansoprazole — Lansoprazole 30 mg, capsules, orally, once daily for up to 6 weeks.
  Other Names: AG-1749
  Arms: Lansoprazole 30 mg QD
Drug: Placebo — TAK-438 placebo-matching tablets, orally, once daily for up to 6 weeks.
  Arms: Lansoprazole 30 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy of TAK-438, once daily (QD), compared to lansoprazole in patients with duodenal ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have endoscopically confirmed duodenal ulcers (mucosal defect with white coating) .At least one ulcer with white coating of 5 mm or larger in size should be observed at baseline (Visit 1).
2. Outpatient (including short inpatient for examination and others)

Exclusion Criteria:

1. Participants with a gastric ulcer which is suspected to be malignant on endoscopy at baseline (Visit 1)
2. Participants with an Acute Duodenal Mucosal Lesion (ADML) on endoscopy at baseline (Visit 1)
3. Participants with a linear ulcer (including scarring) on endoscopy at baseline (Visit 1)
4. Participants with a postoperative ulcer (e.g., Ulcer after EMR/ESD) on endoscopy at baseline (Visit 1)
5. Participants with a gastric ulcer on endoscopy at baseline (Visit 1)
6. Participants with an ulcer for which medical treatment is not indicated (e.g.,perforation, pyloric stenosis, duodenal stenosis, large hemorrhage)
7. Participants who have received endoscopic hemostasis for gastric ulcer within 30 days prior to baseline (Visit 1)
8. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders
9. Participants who have received or who are scheduled to undergo surgery which affects gastric acid secretion (e.g., resection of upper gastrointestinal tract, vagotomy)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Endoscopic Healing Rate of Duodenal Ulcer Over 6 Weeks | 6 weeks
  Endoscopic healing rate : Rate of participants who have endoscopically confirmed all of the white coatings disappeared.

SECONDARY OUTCOMES:
Endoscopic healing Rates of Duodenal Ulcer on Endoscopy over 4 weeks | 4 weeks
Endoscopic healing Rates of Gastric Ulcer on Endoscopy at week 2 | 2 weeks
Change from Baseline in the Incidence of Gastrointestinal Symptoms Associated with Duodenal Ulcer | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (64):
- Japan (64):
  - Toyota-shi, Aichi-ken
  - Kamagaya-shi, Chiba
  - Kisarazu-shi, Chiba
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Kurume-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Tagawa-shi, Fukuoka
  - Yanagawa-shi, Fukuoka
  - Yukuhashi-shi, Fukuoka
  - Sappori-shi, Hokkaido
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Takarazuka-shi, Hyōgo
  - Hitachi-shi, Ibaraki
  - Hitacinaka-shi, Ibaraki
  - Marugame-shi, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Kanoya-shi, Kagoshima-ken
  - Kawasaki-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Yashiro-shi, Kumamoto
  - Kyoto, Kyoto
  - Nagasaki, Nagasaki
  - Sasebo-shi, Nagasaki
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Shimajiri-gun, Okinawa
  - Daito-shi, Osaka
  - Fujiidera-shi, Osaka
  - Hirakata-shi, Osaka
  - Kishiwada-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Suita-shi, Osaka
  - Takatsuki-shi, Osaka
  - Toyonaka-shi, Osaka
  - Saga, Saga-ken
  - Ageo-shi, Saitama
  - Kumagaya-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Ōtsu, Shiga
  - Shizuoka, Shizuoka
  - Ashikaga-shi, Tochigi
  - Otawara-shi, Tochigi
  - Shimotsuga-gun, Tochigi
  - Shimotsuke-shi, Tochigi
  - Tokushima, Tokushima
  - Hachioji-shi, Tokyo
  - Kodaira-shi, Tokyo
  - Kokubunji-shi, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka-shi, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Wakayama, Wakayama
  - Yamagata, Yamagata
  - Shimonoseki-shi, Yamaguchi
  - Kofu, Yamanashi

REFERENCES:
- [Derived] Miwa H, Uedo N, Watari J, Mori Y, Sakurai Y, Takanami Y, Nishimura A, Tatsumi T, Sakaki N. Randomised clinical trial: efficacy and safety of vonoprazan vs. lansoprazole in patients with gastric or duodenal ulcers - results from two phase 3, non-inferiority randomised controlled trials. Aliment Pharmacol Ther. 2017 Jan;45(2):240-252. doi: 10.1111/apt.13876. Epub 2016 Nov 27. PMID 27891632